CLINICAL TRIAL: NCT04943939
Title: Correlation of Electroencephalogram Epileptiform Discharges With Postoperative Delirium During Cardiac Surgery
Brief Title: Correlation of Electroencephalogram With Postoperative Delirium During Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: LN 2021
Record Dates: First submitted 2021-05-20; First posted 2021-06-29 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-06

CONDITIONS: Electroencephalogram; Postoperative Delirium
Keywords: Electroencephalogram; Epileptiform discharges; Postoperative delirium; Cardiac surgery
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to explore characteristic changes of EEG epileptiform discharges in patients under CPB and correlation with POD

DETAILED DESCRIPTION:
Cardiac surgery under cardiopulmonary bypass (CPB) as a result of the surgery itself great trauma and CPB this special process can lead to cerebral hypoperfusion, cerebral ischemia, increased in patients with postoperative neurological complications, the incidence of postoperative cognitive dysfunction can up to 44-53%.Postoperative delirium (POD) is not only increase the incidence of postoperative cognitive dysfunction forward, affect the quality of postoperative recovery and increased hospital costs, also associated with postoperative mortality. Although the clinical use of different drugs and technology improve the POD, but due to the mechanism is still unclear, is still lack of effective control measures. Electroencephalogram (EEG) can measure the cerebral cortex and subcortical local potential activities, to reflect the activities of the neurons in the brain. CPB can cause the abnormal vibration of brain waves, epileptiform discharges is the result of abnormal discharge of brain neurons, which is correlated with the occurrence of cognitive dysfunction.But whether EEG epileptiform discharges is related to the POD is uncertain.While epileptic seizures can be treated with anticonvulsant drugs, so the detection and treatment of early epileptic seizures may have important clinical significance for the occurrence of POD. Therefore, the main purpose of this study is to explore characteristic changes of EEG epileptiform discharges in patients under CPB and correlation with POD, offer the theoretical foundation for delirium early warning and prevention.

ELIGIBILITY:
Inclusion Criteria:

1. ASA II-III;
2. No cognitive impairment was assessed one day before surgery;
3. Patients undergoing elective CPB cardiac surgery(valvular heart surgery and coronary bypass surgery) and signed informed consent.

Exclusion Criteria:

1. Non-CPB surgery, macrovascular surgery, heart transplantation, correction of congenital heart disease;
2. Stroke, schizophrenia, depression, Parkinson's disease, epilepsy or dementia;
3. Inability to communicate with language impairment or major hearing or visual impairment;
4. Liver function child-pugh Grade C, severe liver dysfunction;
5. Severe renal insufficiency requires preoperative renal replacement therapy;
6. A past history of intraoperative knowledge.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cardiac surgery patients
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium after cardiac surgery | The first day after surgery
  Postoperative evaluation delirium occurrence use the The Confusion Assessment Method(CAM) or The Confusion Assessment Method-intensive care unit(CAM-ICU).
Incidence of delirium after cardiac surgery | The second day after surgery
  Postoperative evaluation delirium occurrence use the CAM or CAM-ICU.
Incidence of delirium after cardiac surgery | The third day after surgery
  Postoperative evaluation delirium occurrence use the CAM or CAM-ICU.

SECONDARY OUTCOMES:
Epileptic discharge in electroencephalogram during cardiac surgery | Awake state after entering the operating room (baseline)
  The electroencephalogram (EEG) was collected by Masimo instrument, and the EEG was recognized by the neuroelectrophysiologist
Epileptic discharge in electroencephalogram during cardiac surgery | Start induction of anesthesia until leave the operating room
  The electroencephalogram (EEG) was collected by Masimo instrument, and the EEG was recognized by the neuroelectrophysiologist

CONTACTS AND LOCATIONS:
Overall Officials: Xinli Ni, doctor, Study Chair — General Hospital of Ningxia Medical University
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China